CLINICAL TRIAL: NCT05911243
Title: A Randomized Controlled Trial Testing the Effects of an Acupressure Intervention on Appetite and Weight in Patients With Gastric, Esophageal, and Pancreatic Cancer: A Pilot and Feasibility Study
Brief Title: Feasibility of Auricular Acupressure for Appetite and Weight in Patients With Stage II-IV Gastric, Esophageal, and Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RG1123492; NCI-2023-03942 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1123492 (Other: Fred Hutch/University of Washington Cancer Consortium); 3KL2TR002317 (NIH)
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Acupressure; Practice Guidelines as Topic; Standard of Care; Specimen Handling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (acupressure therapy) (Experimental): Patients undergo auricular acupressure in addition to their usual care on study. Patients also undergo collection of blood samples on study.
  Interventions: Procedure: Acupressure Therapy; Other: Best Practice; Procedure: Biospecimen Collection; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients receive usual care on study. Patients also undergo collection of blood samples on study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Acupressure Therapy — Undergo auricular acupressure
  Other Names: Acupressure; Ischemic Compression
  Arms: Arm I (acupressure therapy)
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This clinical trial evaluates the feasibility and acceptability of acupressure to the ear (auricular) to address appetite and weight in patients with stage II-IV gastric, esophageal, or pancreatic cancer. Cancer anorexia, the abnormal loss of appetite, directly leads to cancer-associated weight loss (cachexia) through malnourishment, reduced caloric intake, treatment side-effects, and other modifiable risk factors. Cachexia prolongs length of hospital stay for patients, negatively impacts treatment tolerance and adherence, and reduces overall patient quality of life. Auricular acupressure is a form of micro-acupuncture that exerts its effect by stimulating the central nervous system using adhesive taped pellets applied to specific locations on the external ear. The use of these pellets to deliver auricular acupressure has been shown to improve pain, fatigue, insomnia, nausea and vomiting, depression, and quality of life in both cancer and non-cancer settings. Auricular acupressure is a safe, inexpensive, and non-invasive approach to addressing cancer-related symptoms and treatment side-effects and may be effective at improving appetite and weight loss in stage II-IV gastric, esophageal, and pancreatic cancer patients.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo auricular acupressure in addition to their usual care on study. Patients also undergo collection of blood samples on study.

ARM II: Patients receive usual care on study. Patients also undergo collection of blood samples on study.

After completion of study treatment, patients in Arm II are followed up at 8 weeks after active treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Stage II-IV gastric, esophageal, or pancreatic cancer
* Appetite score on visual analog scale ≤ 70/100
* At least 60 days of planned systemic treatment, whether already initiated or scheduled to be initiated
* Access to phone and electronic device for study contacts and questionnaires
* Willing and able to attend 4 in-person auricular acupressure treatments at the Fred Hutch South Lake Union Clinic
* Willing and able to perform 4 at-home self-applied treatments of auricular acupressure
* Participants must not have received acupressure or acupuncture for low appetite within last 30 days
* Participants must not be actively using corticosteroids, mirtazapine (Remeron), olanzapine (Zyprexa), or Marinol for appetite stimulation at baseline
* Participants must be able to intake food orally and not require sole or supplemental intravenous nutrition at baseline
* Participants must not have a history of physiological eating disorders (e.g., anorexia nervosa) in the last 3 years
* Participants must not have a current known or diagnosed immunodeficiency
* Participants must have an intact auricular pinna
* Able to understand and willing to sign written informed consent in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accrual (feasibility) | Up to 15 months
  Accrual will be measured by the average rate of participants-per-month enrolled into both groups with the goal of 5 patients/month over a 15-month period.
Retention (feasibility) | Up to 8 weeks
  Retention will be measured by the number of participants who remain in the trial and provide data at the closeout visit.
Intervention adherence (feasibility) | Up to 8 weeks
  Adherence will be measured in the intervention group by the number of applied auricular acupressure treatments, with the total possible being 8.
Intervention fidelity (feasibility) | Up to 8 weeks
  Fidelity will be assessed by study team adherence to symptom query and appropriate ear seed point modifications to the standard protocol and accuracy of seed placement according to photographic analysis.
Acceptability (feasibility) | Up to 16 weeks
  Acceptability will be assessed using a random convenience sample of participants and providers through semi-structured interviews.

SECONDARY OUTCOMES:
Change in appetite | Baseline to week 4
  As measured by the Functional Assessment for Anorexia/Cachexia Treatment Subscale. Analyses will assess change in each outcome as a change from baseline to week 4.
Change in appetite | Baseline to week 8
  As measured by the Functional Assessment for Anorexia/Cachexia Treatment Subscale. Analyses will assess change in each outcome as a change from baseline to week 8.
Change in body weight (kg) | Baseline to week 4
  Analyses will assess change in each outcome as a change from baseline to week 4.
Change in body weight (kg) | Baseline to week 8
  Analyses will assess change in each outcome as a change from baseline to week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Blake Langley, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in published articles after de-identification may be made available upon request (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and ending 36 months after publication of results or study protocol, as requested.
Access Criteria: Researchers and investigators who: 1) provide a methodologically sound proposal to expand on aims in the original, approved proposal; and/or 2) aim to conduct individual, participant-level meta-analyses. Proposals should be directed to blangley@fredhutch.org. To gain access, data requestors will need to sign a data access agreement.